CLINICAL TRIAL: NCT00319956
Title: Trial II of Lung Protection With Azithromycin in the Preterm Infant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hubert Ballard (Other)
Collaborators: American Lung Association (Other)
Responsible Party: Sponsor-Investigator, Hubert Ballard, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 04-0436
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: premature infant; respiratory distress syndrome; mechanical ventilation
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Respiratory Distress Syndrome | interventions — Azithromycin; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin Group (Active Comparator): Group receives azithromycin
  Interventions: Drug: Azithromycin
- Placebo Group (Placebo Comparator): Group receives placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Give 10 mg/kg IV/PO daily for first 7 days, then give 5 mg/kg IV/PO daily for 35 days.
  Other Names: zith, azith
  Arms: Azithromycin Group
Drug: Placebo — vehicle dose given daily, IV/PO, same volume that Azithromycin would be to equal 10 mg/kg for first 7 days, then 5 mg/kg for 5 weeks.
  Other Names: control group
  Arms: Placebo Group

SUMMARY:
The hypothesis of this study is that administration of azithromycin to ventilated premature infants will decrease the incidence and severity of BPD.

The purpose of this study is to determine if Azithromycin treatment is beneficial for prevention of bronchopulmonary dysplasia in preterm infants.

DETAILED DESCRIPTION:
The survival of preterm infants has increased dramatically and has been associated with an increase in BPD. The incidence of BPD among extremely low birthweight infants ranges from 45% to 90%. Development of BPD is associated with both antenatal (maternal chorioamnionitis often due to Ureaplasma is related to BPD) and postnatal complications (oxygen toxicity, barotrauma, late onset infections). These insults appear to lead to an inflammatory response with resultant arrest of normal alveolar and vascular development. Multiple human studies support the role of inflammation in the development of BPD.

Evaluating a medication that could decrease the inflammation in BPD, with minimal side effects, could significantly improve the morbidities of prematurity and the financial burden incurred by parents. Macrolide antibiotics (erythromycin and azithromycin) have been shown to have anti-inflammatory properties that are independent of their antimicrobial properties.

Azithromycin has the potential to decrease the severity of ventilator-induced pulmonary inflammation that is commonly seen in BPD.

ELIGIBILITY:
Inclusion Criteria:

* birthweight less than 1250 grams admitted to UK NICU
* mechanical ventilation within the first 72 hours of life

Exclusion Criteria:

* confirmed sepsis by blood culture
* multiple congenital anomalies or known syndromes
* intrauterine growth retardation with birthweight less than 10%ile for gestational age
* ROM for >7 days

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2004-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hubert O Ballard, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

REFERENCES:
- [Derived] Ballard HO, Shook LA, Bernard P, Anstead MI, Kuhn R, Whitehead V, Grider D, Crawford TN, Hayes D Jr. Use of azithromycin for the prevention of bronchopulmonary dysplasia in preterm infants: a randomized, double-blind, placebo controlled trial. Pediatr Pulmonol. 2011 Feb;46(2):111-8. doi: 10.1002/ppul.21352. Epub 2010 Oct 20. PMID 20963840

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruitment started 9/04 ended 8/08. All subjects were enrolled after admission to NICU. Randomized treatment started within 12 hrs of beginning ventilatory support. If outborn, consent was obtained from parent(s) after phone discussion by the research staff. The consents were faxed, witnessed and brought back by the Transport Team.
Groups:
- Azith Group: Azithromycin : Give 10 mg/kg IV/PO daily for first 7 days, then give 5 mg/kg IV/PO daily for 35 days.
- Placebo Group: D5W : Dose given daily, IV/PO, same volume that Azithromycin would be to equal 10 mg/kg for first 7 days, then 5 mg/kg for 5 weeks.
Period: Overall Study
Arm/Group | Azith Group | Placebo Group
Started | 111 | 109
Completed | 91 | 85
Not Completed | 20 | 24
Not completed — Death | 20 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azith Group | Placebo Group | Total
Number analyzed (Participants) | 111 | 109 | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 111 | 109 | 220
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: gestational age, weeks] | 25.7 (1.5) | 26 (1.6) | 25.85 (1.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 59 | 108
  Male | 62 | 50 | 112
Region of Enrollment [Number; unit: participants]
  United States | 111 | 109 | 220

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Bronchopulmonary Dysplasia (BPD)
Description: comparison of the % Incidence of bronchopulmonary dysplasia (BPD) for the azithromycin vs placebo groups.
Time Frame: diagnosis of BPD at 36wks corrected gestational age
Population: Mortality was 18% in the Azithromycin group and 22% in the Placebo group, thus 91 participants in the Azithromycin group and 85 participants in the Placebo group were analyzed.
Measure: Number; unit: percentage w/ BPD
Arm/Group | Azith Group | Placebo Group
Number analyzed (Participants) | 91 | 85
percentage w/ BPD | 76 | 84
Statistical Analysis 1: Comparison: Azith Group vs Placebo Group; Test type: Superiority; p = 0.20, Chi-squared

2. Other Pre Specified Outcome: Postnatal Steroid Use
Description: Steroids will be provided as needed based on Standard of Care. Data are presented as the percent of participants that received steroids between birth and discharge from the NICU.
Time Frame: Duration of NICU stay, up to 16 weeks, average stay is about 10 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Azith Group | Placebo Group
Number analyzed (Participants) | 111 | 109
percentage of participants | 18 | 22

3. Other Pre Specified Outcome: Number of Days on Mechanical Ventilation
Description: Participants will be placed on mechanical ventilation as necessary based on standard of care. Data are presented as the percent of participants in each group receiving mechanical ventilation.
Time Frame: Duration of NICU stay, up to 16 weeks, average stay is about 10 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Azith Group | Placebo Group
Number analyzed (Participants) | 111 | 109
days | 28 (26) | 26 (26)

4. Other Pre Specified Outcome: Participant Mortality
Description: Data will be collected on the number of participants that did not survive to discharge from the NICU. Data are presented as the percent of participants that did not survive.
Time Frame: Duration of NICU stay, up to 16 weeks, average stay is about 10 weeks
Measure: Number; unit: percentage of mortality
Arm/Group | Azith Group | Placebo Group
Number analyzed (Participants) | 111 | 109
percentage of mortality | 18 | 22

ADVERSE EVENTS:
Time Frame: 1 year.
Arm/Group | Azith Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 20/111 | 24/109
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/109
Other Adverse Events (participants affected / at risk) | 0/111 | 0/109

LIMITATIONS AND CAVEATS:
The number of participants for this study was quite small. A large scale trial is required to draw any conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes